CLINICAL TRIAL: NCT02986529
Title: A Double-blind, Randomized, Three-period, Three-way Crossover Design, Placebo Controlled Single Dose Study to Assess the Bioavailability of Sodium Oligo-mannurarate (GV-971) Capsule 150 mg, 300mg, 450mg in Healthy Chinese Male Subjects
Brief Title: A Study to Assess the Bioavailability of Oral Sodium Oligo-mannurarate (GV-971) in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Greenvalley Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRC-C1503
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2017-12

CONDITIONS: Bioavailability
MeSH Terms: interventions — GV-971

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GV-971 150mg/capsule (Active Comparator): 900mg, oral
  Interventions: Drug: GV-971
- GV-971 300mg/capsule (Experimental): 900mg, oral
  Interventions: Drug: GV-971
- GV-971 450mg/capsule (Experimental): 900mg, oral
  Interventions: Drug: GV-971
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: GV-971
  Other Names: Sodium Oligo-mannurarate
  Arms: GV-971 150mg/capsule; GV-971 300mg/capsule; GV-971 450mg/capsule
Drug: Placebos
  Arms: Placebo

SUMMARY:
To evaluate the Bioavailability for GV-971 capsules of 150 mg, 300mg, and 450mg after administration of single oral doses of 900mg in healthy Male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects;
2. Age：≥18 and ≤45 on the date signing informed consent
3. Body mass index (BMI): 18-25 kg/m2 and the weight ≥50 kg；
4. Subjects are able to understand the study procedures and methods, and willing to strictly comply with the protocol and give written informed consent.

Exclusion Criteria:

A subject will be excluded if the answer to any of the following criteria is "yes":：

1. Clinically significant abnormalities in physical examination and laboratory test results or 12-lead ECG, etc. in screening;
2. Clinically significant abnormalities in Chest X-ray or abdominal B-ultrasound examination
3. Positive serology screen for Hepatitis B( HBsAg), Hepatitis C(HCV), HIV and USR unheated serum reagin test.
4. Smoking more than 10 cigarettes a day, drugs or alcohol abuse within 6 months prior to screening
5. Participation in any investigational drug or medical instrument study within 3months prior to screening, participation in 3 and more than 3 drug tests in a recent year;
6. Serious infection, trauma and major surgery within 4weeks prior to screening;
7. Blood donation of ≥400 mL or severe blood lose and the volume of blood loss ≥400 mL within 4 weeks prior to screening, receiving blood transfusion treatment within 8 weeks prior to screening ;
8. Use of any prescription medicine or herbal remedy, over the counter medication or dietary supplements such as vitamin, calcium within 2 weeks prior to screening.
9. Use of heparin, alginic sodium diester , mannose ester within 4 weeks prior to screening；
10. Vegetarian or person with dietary restrictions
11. Subjects able to father a child are unwilling to use highly effective physical form of birth control from the trial period until 3 months after the completion of study.
12. With diseases which could impact on the absorption, distribution, metabolism and excretion (ADME) of study drugs or protocol adherence in the opinion of the investigator (such medical disorder/disease may relate to ccardiovascular, liver, kidney, digestive, immune, blood, endocrine, metabolic, cancer, neuropsychiatric,etc );
13. Subjects may be allergic to GV-971 in the opinion of the investigator.
14. Any other reasons that the subject is not eligible for participation in the study in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02-24 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Cmax - maximum observed concentration, is obtained directly from the plasma concentration curve | 3 days
AUC0-last-the area under the concentration-time curve from zero to the time of the last measurable concentration; computed using the linear trapezoidal rule | 3 days
AUC0-∞-the area under the concentration-time curve from zero to the infinity, computed as AUC0-∞=AUC0-last+Clast/λz (λz is the terminal phase rate constant) | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Phase-I Clinical Research Unit at Shanghai Xuhui Center hospital, Shanghai, Shanghai Municipality, China